CLINICAL TRIAL: NCT05871853
Title: Getting the Benefits From the Beginning. Improving Breastfeeding Support for Families at Risk of Breastfeeding Difficulties
Brief Title: Get the Benefits From the Start. Improving Breastfeeding
Status: Recruiting | Type: Observational
Sponsor: Slagelse Hospital (Other)
Collaborators: Center for Clinical Research and Prevention (Network); Region Zealand (Other); Steno Diabetes Center Sjaelland (Other Government)
Responsible Party: Principal Investigator, Annemi Lyng Frandsen, Ph. D. Student, Slagelse Hospital
Other Study IDs: REG-094-2022
Record Dates: First submitted 2023-05-15; First posted 2023-05-23 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; Infant; Newborn; Post-natal Care
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-implementation group: Women delivering during an eight month period, before the intervention is implemented.
- Post-implementation group: Women delivering during an eight month period, after the intervention is implemented.
  Interventions: Behavioral: Improved breastfeeding support

INTERVENTIONS:
Behavioral: Improved breastfeeding support — Cross-sectoral intervention to improve breastfeeding support among women giving birth at Slagelse Hospital, Region Zealand, Denmark
  Groups: Post-implementation group

SUMMARY:
Breastfeeding is beneficial for the physical and mental health of mothers and infants alike.

Most new mothers in Denmark intend to breastfeed, however, a substantial proportion do not succeed to breastfeed as intended.

In Region Zealand, few women breastfeed than in the rest of Denmark in which may be related to a higher proportion of women being overweight, having socio-economic constraints and a low educational level, all associated with breastfeeding difficulties. There is limited knowledge on how to deliver a tailored support aimed at families at high risk of breastfeeding difficulties in a high-income country.

We plan to conduct a study aiming to strengthen breastfeeding support to families at risk of breastfeeding difficulties, delivering at Slagelse Hospital, across healthcare sectors, including obstetric and neonatal departments, primary care and civil society.

The study aims to develop, implement, and evaluate a supportive breastfeeding intervention with specific focus on families at high risk of complicated breastfeeding and early breastfeeding cessation - a prospective cohort study in Region Zealand, Denmark.

Potentially, results can help reducing inequality in health thus more families achieve exclusive breastfeeding and gain health benefits from breastfeeding

DETAILED DESCRIPTION:
Background. Breastfeeding is a tailored nutrition for newborn infants in their first years. Breastfeeding has short and long-term positive health effects on both mothers and infants.

For infants, breastfeeding has a protective effect against sudden infant death, respiratory, gastrointestinal and ear infections, obesity, diabetes and childhood leukemia. Breastfeeding also benefits the infant's cognitive development. Studies have found that breastfeeding positively affects the infant's cognitive abilities and IQ. For premature infants, mothers' own milk also protects against the potentially life-threatening disease necrotizing enterocolitis as well as reducing the risk of retinopathy of prematurity for very preterm infants.

For mothers, breastfeeding carries a reduced risk of type 2 diabetes, breast- and ovarian cancer and reduce the risk of cardiovascular disease and benefits the mothers because it may reduce depression and stress. Furthermore, breastfeeding may increase a secure mother-infant attachment, and improve the mother's emotional response to the infant, proportionally with the duration of breastfeeding.

The World Health Organization(WHO) recommends exclusive breastfeeding for six months and partially for two years or longer and has set a goal of optimizing breastfeeding in 2025. Danish Health Authorities also recommend exclusive breastfeeding for six months and partially for one year or longer.

Internationally breastfeeding rates and duration has declined and Denmark is no exception. Breastfeeding has a social barrier both in the early phase of initiation and in the first months, in low-income as well as in high-income countries. We know that breastfeeding follows a pattern of inequalities, and women with less education and low socio-economic status are less likely to exclusively breastfeed.

Declining rates of breastfeeding are a growing problem, as exclusive breastfeeding has decreased over the last decade in all Danish regions. Region Zealand is one of the regions with the lowest rate of exclusive breastfeeding when the infant is four months old compared to the rest of Denmark. Even though Denmark has a relatively well developed health care system with (at least formal) equal access to health services, inequality in health is growing, especially in Region Zealand.

Certain factors are known to be associated with difficulties in initiating and sustaining breastfeeding. These include maternal overweight, gestational diabetes, delivery by cesarean section, admission of the infant to Neonatal Intensive Care Unit (NICU) due to being small, premature or sick, as well as breastfeeding problems with a previous child, previous operations on the breast, social and economic constraints and psychosocial problems for the mother.

In Denmark, we have guidelines for breastfeeding counselling after uncomplicated birth. We know that early interventions will change the trajectory of non-infectious diseases. We lack, however, knowledge on how to offer differentiated care for breastfeeding mother and infant dyads with risk factors for complicated breastfeeding, including how we can improve collaboration with healthcare visitors in the municipalities to make the best transition from hospital to home. We do not have differentiated programs so we help the families who need help the most.

Purpose and hypotheses. This study aims to develop, implement and assess the effect of cross-sectoral cooperation aiming to support breastfeeding in families who give birth at Slagelse Hospital and who are at high risk of complicated breastfeeding. We intend to set up a new service where we provide families at high risk of complicated breastfeeding, with differentiated, practical counselling based on the family's needs, and evidence-based knowledge.

Our hypothesis is that an early differentiated and locally adapted intervention will increase the initiation rate and duration of breastfeeding among women delivering at Slagelse Hospital.

The study is an independent part of an initiative at Slagelse Hospital, Region Zealand, aiming to reduce inequality in health among children.

The study design is a clinical prospective observational cohort study: The development, implementation, and evaluation of a supportive breastfeeding intervention with specific focus on families at high risk of complicated breastfeeding and early breastfeeding cessation - a prospective cohort study in Region Zealand, Denmark.

Aim. To develop, implement and evaluate a locally adapted and differentiated breastfeeding-counselling model, focusing especially on families at risk of experiencing breastfeeding difficulties, and therefore most likely to benefit from health-promoting efforts like breastfeeding support.

Research question. Will the implementation of a locally adapted intervention aimed at supporting families at high risk of complicated breastfeeding outcomes lead to an increase in the proportion of exclusively breastfed children at four months of age when compared to a cohort born before the intervention?

Study design. In a prospective, observational design, we will follow families delivering during eight months following the implementation of the intervention and compare to a control group of families delivering during eight months before the intervention.

Intervention. The intervention is a complex process and we will therefore use a theoretical framework for complex interventions developed by the Medical Research Council, as a sustainable effort for breastfeeding, requires collaboration across sectors, the involvement of various health professions and the involvement of users and stakeholders from the local community.

The exact design of the intervention will therefore be determined according to the results of this process.

However, the intervention is likely to include components described in the WHO's Baby Friendly Hospital Initiative (BFHI) and neonatal BFHI:

We plan to stratify the intervention by identifying women at risk either at prenatal consultations during pregnancy, or at birth:

1. Women with low risk factors will be given the care described in Danish National Guideline for initiation of breastfeeding after an uncomplicated birth
2. Women with a moderate risk will be offered a seven day program with easy contact to the maternity ward as described by the Danish Health Authorities in the early postpartum period
3. Women with high risk will be offered a tailored intervention with an easy access to qualified breastfeeding counselling. This service will be planned in co-creation with peer support groups from the organization "Forældre og Fødsel", midwives and nurses at the Slagelse hospital maternity ward, nurses at the Slagelse hospital neonatal ward, and health visitors from three municipalities in Region Zealand.

Although the intervention has a specific focus on those in the highest risk, it may also improve the care given to families at lower risk of breastfeeding complication by raising general awareness and improving the knowledge among health care workers.

Materials and methods. We will perform a prospective observational cohort study, following families giving birth during the eight months before the intervention (pre-cohort), compared to a cohort of families giving birth during eight months after the intervention is implemented (post-cohort). Children born during a pilot phase of 4 months between the pre-cohort and the complete implementation of the intervention will not be included in the data collection.

Participants. Primarily the intervention aims at families in a target group of families at high risk of complicated breastfeeding; however, as the intervention may also include a general change of culture and attitude, as well as a general improved training among health staff, it may potentially benefit all families. We will therefore collect data from all families delivering at the hospital, including families in the target group, and from low-risk families delivering at the hospital who give consent to participate in the study (collect data).

Data collection. Data will be collected on all consenting families giving birth at Slagelse Hospital in the period of eight months before the intervention, and one year after. Consent to collect and store patient data will be obtained from families at inclusion.

Data on primary and secondary outcomes will be collected through electronic questionnaires after discharge. If the families do not fill out (in) the questionnaires themselves, they will be contacted by telephone.

Power and sample size estimation. It is assumed that 50% of all women currently breastfeed their child for four months based on the Danish Child Database(18). Showing an increase after the intervention to 57% with a power of 80% and alpha of 0.05 requires that we include 796 families in the control and intervention cohort. This is estimated to be achievable as there are approximately 1,800 births annually Slagelse Hospital. This means that in 8 months there are approximately 1,200 women giving birth, of which 80% are expected to give consent for data collection, corresponding to 960 families.

ELIGIBILITY:
Inclusion Criteria:

* All women giving birth at Slagelse Hospital and their infants during the study period
* Age at 15 years and above

Exclusion Criteria:

* families with a planned placement of the infant in a fostercare

Ages: 15 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women giving birth as well as their infants For twins and multiples; only the first born.
Study Population: Women giving birth at Slagelse Hospital and their actual infant
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of mother's self-reporting exclusive breastfeeding | 4 month postpartum
  Mothers who are exclusive breastfeeding in the post-implementation group, compared to the pre-implementation group (n/% of total).
  Exclusive breastfeeding is defined as exclusive fed at the breast after discharge from hospital. This means, that in addition to breastfeeding, supplements with water and similar and/or a or a maximum of one meal of breastmilk substitute or mothers expressed breastmilk per week.

SECONDARY OUTCOMES:
Duration of exclusive breastfeeding | 0-12 month
  Duration of mothers' self-reporting exclusive breastfeeding in the post-implementation group, compared to the pre-implementation group (days, median with IQR).
Duration of any breastfeeding | 0-12 month
  Duration of mothers' self-reporting any breastfeeding in the post-implementation group, compared to the pre-implementation group (days, median with IQR).
Rate of exclusive breastfeeding reported by the home-visiting nurse | 4 months
  Mothers who are exclusive breastfeeding in the post-implementation group, compared to the pre-implementation group. Reported from the Danish National cross-sectoral database at (n/% of total).
Any admission of the infant | 0-12 month
  Any admission of the infant to hospital or referral to a pediatric outpatient clinic compared with any breastfeeding in the post-implementation group, compared to the pre-implementation group (n/% of total).
Mothers self-reported well-being | Third trimester, 14 days, 1 month, 4 month, 6 month after birth
  Mother's self-reported well-being measured by WHO 5 in the post-implementation group compared to the pre-implementation group. (mean (SD) cut off ><50 indicating clinical depression)
Infant well-being as reported by the mother | 4 month
  Mother's selfreported infant health related quality of life (TANDI) in the post-implementation group compared to the pre-implementation group at age of four month.
Proportion of children sucking at the breast within the first hour of life | 1 hour of life
  The proportion of children sucking at the breast within the first hour of life, in the post-implementation group compared to the pre-implementation group. Reported by the mother at 14 days postpartum (n/%total).
Time spend skin-to-skin on 14th day of life | Day 13
  Time (hours) spend skin-to-skin on the previous day as reported by the mother at 14 days postpartum in the post-implementation group compared to the pre-implementation group (hours/24 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Annemi L Frandsen, MSA, Principal Investigator — Børne- og Ungeafdelingen, Slagelse Sygehus
Locations (1):
- Slagelse Hospital, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
We plan to upload anonymized data to a data repository